CLINICAL TRIAL: NCT01204281
Title: High-assistance Proportional Assist Ventilation (PAV) vs. Assist-Control Ventilation (ACV) in Early Stage of Critically Ill Patients
Brief Title: Proportional Assist Ventilation (PAV) in Early Stage of Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Rafael Fernandez, Head of Intensive Care Department, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIC 10-48
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Respiratory Failure; Mechanical Ventilation
Keywords: Proportional Assist Ventilation plus; Acute respiratory failure; Mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Interactive Ventilatory Support; Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High assistance PAV+ (Experimental): Ventilatory support performed by PAV at 80% assistance (PB 840-plus) FiO2 and PEEP according to routine practice
  Interventions: Other: Mechanical ventilation mode (PAV+ vs. ACV)
- Assist-control ventilation (Active Comparator): Tidal volume, FiO2 and PEEP set according to routine practice
  Interventions: Other: Mechanical ventilation mode (PAV+ vs. ACV)

INTERVENTIONS:
Other: Mechanical ventilation mode (PAV+ vs. ACV) — Compare two ventilatory modes in the acute phase of illness
  Other Names: Proportional Assist ventilation (PAV+); Assist Control ventilation; Critically ill patients; Mechanical ventilation

SUMMARY:
To evaluate the effectiveness of high assistance proportional assist ventilation (PAV+) (objective 80% gain) as main ventilatory support in early stage of critically ill patients in comparison with standard volume-assist control ventilation (ACV).

DETAILED DESCRIPTION:
The goal of this proposal is to apply PAV+ as routine ventilatory mode in the early stage of critically ill patients, taking advantages of spontaneous breathing and better patient-ventilator interaction.

The standard treatment in patients with acute respiratory failure is mechanical ventilation in control-mode for the first days of acute illness. This procedure is usually associated with patient-ventilator dyssynchrony, higher needs of sedation and/or relaxation, muscle atrophy, etc. PAV + is a new ventilatory mode that applies pressure in proportion to spontaneous patient inspiratory effort allowing better adaptation to changes in internal homeostasis.

Up to now, several reports compare PAV with assisted modes as a feasible alternative only in the weaning phase. However, PAV is able to unload patient effort in different levels, suggesting that high-assistance PAV (about 80%) could be comparable with assist-control modes in terms of respiratory muscles unload.

Whether PAV is as effective as traditional ACV in terms of ventilation muscle unload in the acute phase of illness has not been established and we aim to address this question.

We plan to prospectively enroll patients on mechanical ventilation early at ICU admission, and to ventilate them randomly under ACV (volume-assist control ventilation) or PAV+ (beginning with 80% if possible). We will evaluate length of mechanical ventilation, sedation requirements and respiratory-hemodynamic variables from the very beginning and until attending clinicians decide that patients are ready to be weaned.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Anticipated MV > 24 hours
* Availability of informed consent from patient or next of kin
* Ventilation parameters measured under PAV+ 80% gain:

PaO2/FiO2 >100 RPAV <10 cm H2O/l/s CPAV > 30 ml/cm H2O WOBTOT <1.5 J/l VE <18 l/min

Exclusion Criteria:

* Patients on moribund state or with life-sustaining therapy withholding decision.
* Patients with unstable respiratory/hemodynamic state, PaO2/FiO2 <100, Dopamine >15 microg/Kg/min or epinephrine >0.1 microg/kg/min.
* Pregnancy.
* Air leak.
* Patients needing deep sedation or muscle paralysis
* Patients needing hyperventilation (brain trauma).
* Patients with severe muscle weakness.
* Recruitment maneuvers or prone position.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Length of mechanical ventilation | 28 days
  Reduction of mechanical ventilation days when ventilated with high assistance PAV+ compared with ACV.

SECONDARY OUTCOMES:
Non-inferiority of PAV+ compared to ACV in terms of gas exchange | 28 days
  Non-inferiority of high assistance PAV+ compared to ACV in terms of gas exchange
Noninferiority of PAV in short term complications | 28 days
  Similar incidence in the complications composite outcome (barotrauma, ARDS, atelectasis and pneumonia)
Noninferiority of PAV in weaning success | 28 days
  Similar rate of weaning success defined as the composite end-point: time to resume spontaneous ventilation, rate of extubation success, need for non invasive ventilation (NIV) as rescue therapy, and reintubation rate.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Fernandez, M.D., Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa
Locations (1):
- Intensive Care Unit. Xarxa assistencial Althaia., Manresa, Catalonia, Spain

REFERENCES:
- [Result] Grasso S, Puntillo F, Mascia L, Ancona G, Fiore T, Bruno F, Slutsky AS, Ranieri VM. Compensation for increase in respiratory workload during mechanical ventilation. Pressure-support versus proportional-assist ventilation. Am J Respir Crit Care Med. 2000 Mar;161(3 Pt 1):819-26. doi: 10.1164/ajrccm.161.3.9902065. PMID 10712328
- [Result] Georgopoulos, D., Plataki, M., Prinianakis, G., Kondili, E., Current status of proportional assist ventilation. International journal of Intensive Care, 2007. Autumn: p. 19-26.
- [Result] Delgado M, Zavala E, Tomas R, Fernandez R. "Feasibility of proportional assist ventilation as routine ventilatory support in intensive care patients". Intensive Care Med 2009; 35; Suppl 1: S125
- [Result] Putensen C, Muders T, Varelmann D, Wrigge H. The impact of spontaneous breathing during mechanical ventilation. Curr Opin Crit Care. 2006 Feb;12(1):13-8. doi: 10.1097/01.ccx.0000198994.37319.60. PMID 16394778
- [Result] Younes M. Proportional-assist ventilation. In: Tobin MJ, editor. Principles and practice of mechanical ventilation. Illinois: McGraw-Hill; 2006. p. 335-64.